CLINICAL TRIAL: NCT01796795
Title: A Double-blind, Randomized, Vehicle-controlled, Parallel-group, Phase II Dose-ranging Study to Evaluate the Efficacy and Safety of SR-T100 Gel in Common Warts (CW) Patients.
Brief Title: Efficacy and Safety of SR-T100 Gel in Common Warts (CW) Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Budget issue.
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GESRTCWA
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Common Wart
Keywords: common wart; verruca vulgaris
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- vehicle gel (Placebo Comparator): The vehicle gel will be applied in appropriate amount evenly and gently in a thin-layer of gel by finger, not to exceed 0.2 g per administration (approximately 2 cm gel squeezed in length). Each dose of study drug is applied on the target lesion(s) and covered with an occlusive dressing for the entire day.
  Interventions: Drug: Vehicle gel
- SR-T100 gel with 1.0% of SM (Active Comparator): SR-T100 contains 1.0% SM. The gel will be applied in appropriate amount evenly and gently in a thin-layer of gel by finger, not to exceed 0.2 g per administration (approximately 2 cm gel squeezed in length). Each dose of study drug is applied on the target lesion(s) and covered with an occlusive dressing for the entire day.
  Interventions: Drug: SR-T100 gel with 1.0% of SM
- SR-T100 gel with 2.3% of SM (Active Comparator): SR-T100 contains 2.3%SM. The gel will be applied in appropriate amount evenly and gently in a thin-layer of gel by finger, not to exceed 0.2 g per administration (approximately 2 cm gel squeezed in length). Each dose of study drug is applied on the target lesion(s) and covered with an occlusive dressing for the entire day.
  Interventions: Drug: SR-T100 gel with 2.3% of SM

INTERVENTIONS:
Drug: Vehicle gel — Topical application on the target lesion(s)once daily with occlusive dressing; a maximum of 3 times of administration of gel without exceeding 0.2 g per administration.
  Arms: vehicle gel
Drug: SR-T100 gel with 1.0% of SM — Topical application on the target lesion(s)once daily with occlusive dressing; a maximum of 3 times of administration of gel without exceeding 0.2 g per administration.
  Arms: SR-T100 gel with 1.0% of SM
Drug: SR-T100 gel with 2.3% of SM — Topical application on the target lesion(s)once daily with occlusive dressing; a maximum of 3 times of administration of gel without exceeding 0.2 g per administration.
  Arms: SR-T100 gel with 2.3% of SM

SUMMARY:
This phase II study is to evaluate the efficacy of SR-T100 gel in complete clearance of target warts at different concentrations (1.0% and 2.3% of SM in Solanum undatum plant extract) in patients with CW.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 17 years old.
2. The diagnosis of CW is based on visual inspection by an experienced dermatologist.
3. Patient is selected ≤ 5 CW lesions; each of the target lesion(s) needs to be ≤ 15 mm in diameter. For patient with only 1 selected lesion, the size of target lesion needs to be measuring 2 to 15 mm in diameter.
4. Patient agrees to apply the study medication on target CW lesion(s) with an occlusive dressing for at least 20 hours per day.
5. Patient or the legally acceptable representative of patient under 20 years of age, is willing and able to provide written informed consent.
6. Patient agrees not to use wart-removing product/modality (prescription or over-the-counter) other than the study product during the course of the study; and is willing to refrain from using cosmetics or other topical products in the treatment area for the duration of the study.
7. Any non-target CW receiving wart-removing procedures including cryotherapy and surgical therapy should be at least 5 cm apart from the target lesions.
8. Patient is free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk to the patient.
9. Patient is judged to be in good health based upon the results of physical examinations (PEs), medical history, and safety laboratory tests.
10. Patient in good general health condition (performance status ≤ 2 Eastern Cooperative Oncology Group (ECOG)).
11. Patient agrees to be photographed of the CW target lesion(s) and used of such data as part of the study package.
12. Female patient of childbearing potential should have a negative urine or serum pregnancy test at Screening day, and is willing to use effective contraception during the study.

Exclusion Criteria:

1. The treatment area is located in any of the following areas: the eye area (including eyelids), lips, mouth cavity, nasal cavity,inner ear, soles of the feet, underneath the nails, and the anogenital area.
2. Patient had participated in a clinical study within 30 days prior to the Randomization visit, or is currently participating in another clinical study.
3. Patient had used any wart-removing product/modality in the treatment area within 30 days prior to the Randomization visit or received cryotherapy in the treatment area within 60 days prior to the Randomization visit.
4. Patient who has immune-compromised conditions, have required or will require systemic intake of immunosuppressive or immunomodulatory medication (oral or parental corticosteroids are included) within 30 days prior to the Randomization visit or during the course of the study. Routine use of inhaled or intranasal corticosteroids during the study is allowed.
5. Patient has clinically significant or unstable medical conditions (psychologically and physically) in any of the following listed situations:

   1. Clinically significant peripheral vascular disease based on medical history.
   2. Current uncontrolled infection, current skin infections and/or skin disorder in the treatment area other than CW and/or in the area surrounding the warts that may confound or affect study assessment procedure of the study endpoints.
   3. Chronic or acute medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk (including human immunodeficiency virus, systemic lupus erythematosis, active viral hepatitis, etc.).
6. Patient is pregnant, plan to become pregnant, or is breastfeeding.
7. Patient has a history of allergy or sensitivity to Solanum undatum plant extract, SM, or SR-T100 gel excipients including carbomer, propylene glycol, and triethanolamine.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2030-09 (Estimated); Primary Completion 2033-04 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Total clearance rate of treated CW | 16 weeks

SECONDARY OUTCOMES:
Proportion of patient with at least 75% reduction in CW lesion counts | 16 weeks
Proportion of patient with at least 50% reduction in lesion size (volume) | 16 weeks
Mean of percent reduction in CW lesion counts from individual patient by visit | 16 weeks
Mean of percent reduction in CW lesion size from individual patient by visit | 16 weeks
CW recurrence rate | 28 weeks
Time to complete clearance | 16 weeks
Percent reduction for pooled lesion counts by visit | 16 weeks
Safety: evaluate the changes occurring from baseline (Randomization visit) to EOT visit. | 28 weeks
  including PE, vital sign, lab. test, local skin reaction, and adverse event, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kou-Wha Kuo, Ph.D, Study Director — G&E Herbal Biotechnology Co., LTD; Hamm-Ming Sheu, MD, Principal Investigator — National Cheng-Kung University Hospital